CLINICAL TRIAL: NCT03787251
Title: Randomized, Open, Positive Drug Control, Multicenter Clinical Study of Second-line Treatment of Postoperative Recurrence and Metastasis of Esophageal Squamous Cell Carcinoma With Chemotherapy in Patients Treated With Apatinib Mesylate
Brief Title: A Study of Second-line Treatment of Postoperative Recurrence and Metastasis of Esophageal Cancer Treated With Apatinib
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: In China, apatinib has been approved as an indication drug for esophageal squamous cell carcinoma, which makes it very difficult for our clinical trial to enroll patients. We regret that we failed to implement the design as planned.
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Wei Ren, Deputy Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nanjing Drum Tower Hospital
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2019-01

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): It is recommended that the initial dose of apatinib is 500mg po qd. Adjust the dose to 750mg po qd or maintain the original dose according to the patient's medication response for about 2 weeks. If there is grade III or above, or grade II and above non-hematologic toxicity, allow the dose to be lowered 2 times.
  Interventions: Drug: Apatinib
- Control group (Active Comparator): The chemotherapeutic drug chosen by the investigator (if not used in the previous treatment regimen, it cannot be selected).
  The choice of chemotherapy regimen is based on the medication habits of the drug delivery doctor and the specific circumstances of the patient.
  In addition, the following regimens may be selected as monotherapy or combination: docetaxel 60-75 mg/m2d1 q3w; irinotecan 150-180 mg/m2 d1 q2w until disease progression or patient decease. If the adverse event grade 3 and above Or non-hematologic toxicity of grade II and above appeared, allowing the dose to be lowered twice.
  Interventions: Drug: The chemotherapeutic drug chosen by the investigator.

INTERVENTIONS:
Drug: Apatinib — It is recommended that the initial dose of apatinib is 500mg po qd. Adjust the dose to 750mg po qd or maintain the original dose according to the patient's medication response for about 2 weeks. If there is grade III or above, or grade II and above non-hematologic toxicity, allow the dose to be lowered 2 times.
  Arms: experimental group
Drug: The chemotherapeutic drug chosen by the investigator. — The choice of chemotherapy regimen is based on the medication habits of the drug delivery doctor and the specific circumstances of the patient.
  In addition, the following regimens may be selected as monotherapy or combination: docetaxel 60-75 mg/m2d1 q3w; irinotecan 150-180 mg/m2 d1 q2w until disease progression or patient death. If grade 3 and above or non-hematologic toxicity of grade II and above adverse event appeared, allowing the dose to be lowered twice.
  Arms: Control group

SUMMARY:
A study of second-line treatment of postoperative recurrence and metastasis of esophageal squamous cell carcinoma after chemotherapy with apatinib mesylate

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center, phase II clinical trial initiated by a investigator to observe and evaluate the efficacy of apatinib in the treatment of patients with failed first-line treatment after recurrence and metastasis of esophageal squamous cell carcinoma. Effectiveness and security.

ELIGIBILITY:
Inclusion Criteria:

* Pathological/histological diagnosis of esophageal squamous cell carcinoma; and at least one measurable lesion according to RECIST criteria (version 1.1);
* Patients who have undergone radical resection of esophageal cancer and who have failed after first-line systemic chemotherapy (which may include platinum, taxane or fluorouracil) after recurrence (recurrence of postoperative adjuvant chemotherapy within 6 months) Considered as first-line treatment, and the same progress in the field of radiation can be seen as recurrence;
* Age: 18-75 years old; both men and women;
* ECOG PS Rating: 0-1 points;
* Estimated survival period ≥ 3 months;
* ≥ 4 weeks from the last cytotoxic drug;
* The main organs function normally, that is, meet the following criteria:

  * Blood routine examination:

    * HB≥90 g/L; (no blood transfusion within 14 days)
    * ANC ≥ 1.5 × 109 / L;
    * PLT ≥ 80 × 109 / L;
  * Biochemical examinations must meet the following criteria:

    * ALT and AST < 2.5 ULN; if there is liver metastasis, ALT and AST < 5 ULN;
    * TBIL ≤ 1.5ULN;
    * Plasma Cr≤1.5ULN or creatinine clearance (CCr)≥60ml/min
* Subjects volunteered to participate in the study, signed informed consent, and were well-adhered to follow-up.
* Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months of the end of the study; negative serum or urine pregnancy tests within seven days prior to study enrollment And must be non-lactating patients; males should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* Those who have used anti-tumor angiogenesis drugs to treat failure;
* Patients with residual esophagus, residual stomach or anastomotic recurrence;
* Unable to swallow, chronic diarrhea and intestinal obstruction, which obviously affect the taking and absorption of drugs;
* Patients with brain metastases with symptoms or symptoms controlled for less than 3 months;
* Long-term unhealed wounds and fractures;
* Have clear gastrointestinal bleeding concerns (such as local active ulcer lesions, fecal occult blood above ++), history of gastrointestinal bleeding within 6 months; coagulation abnormalities (PT>16 s, APTT>43 s, TT>21 s, Fbg< 2 g/L), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
* Overactive/venous thrombosis occurred within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism;
* Imaging shows that the tumor has invaded the important perivascular circumference or that the patient is likely to invade the important blood vessels during the follow-up study and cause fatal bleeding.
* Persons with a history of psychotropic substance abuse who are unable to resolve or have a mental disorder;
* Participated in other clinical trials of anti-tumor drugs within four weeks;
* Have a history of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
* According to the investigator's judgment, there are serious concomitant illnesses that compromise the safety of the patient or affect the patient's completion of the study.
* Patients with any severe and/or uncontrolled diseases, including:

  * Blood pressure control is unreasonable (retraction pressure >150mmHg, diastolic pressure >100mmHg) Patients: I have myocardial ischemia or myocardial infarction above grade I, arrhythmia (including QT interval >440ms) and grade I cardiac insufficiency;
  * Active or uncontrolled serious infections;
  * Liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis;
  * Poor diabetes control (fasting blood glucose FBG>10mmol/L);
  * Urine routine indicates urinary protein >++, and confirmed 24-hour urine protein quantitation >1.0g.
* The investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | One year from admission
  progression-free survival

SECONDARY OUTCOMES:
OS | One year from admission
  Overall Survival
DCR | One year from admission
  disease control rate
ORR | One year from admission
  Objective Response Rate